CLINICAL TRIAL: NCT02936440
Title: Assessment of Hydration Status Using Bioelectrical Impedance Vector Analysis in Critical Patients With Acute Kidney Injury
Brief Title: Assessment of Hydration Status Using Bioelectrical Impedance Vector Analysis
Status: Completed | Type: Observational
Sponsor: Catholic University of Pelotas (Other)
Responsible Party: Principal Investigator, Maria Cristina Gonzalez, Full Professor, Catholic University of Pelotas
Other Study IDs: 2009/79
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Acute Kidney Injury; Critical Illness
Keywords: acute kidney injury; intensive care unit; bioelectrical impedance analysis
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critical patients with AKI: Critical patients with AKI will be followed up to 12 weeks after diagnosis

SUMMARY:
The state of hyperhydration in critically ill patients with acute kidney injury (AKI) is associated with increased mortality. Bioelectrical impedance vector analysis (BIVA) appears to be a viable method to access the fluid status of critical patients but has never been evaluated in critical patients with AKI. The objective of this study is to evaluate the hydration status using BIVA in critical patients under intensive care at the time of AKI diagnosis and to correlate this measurement with mortality. A sample of 224 patients with AKI will be evaluated by BIVA and followed until they are discharged or death in intensive care unit and the BIVA vectors will be analysed to define differences in hydration characteristics from each group.

DETAILED DESCRIPTION:
Patients admitted to Intensive Care Unit (ICU) will be assessed by BIVA at the moment of the AKI diagnosis. They will be followed up to 12 weeks, until hospital discharge or death. The association between survival and hydration status, as assessed by BIVA in the first AKI day, will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years who developed acute kidney injury after admission in Intensive Care Unit

Exclusion Criteria:

* Chronic kidney injury, dialysis-dependent chronic kidney injury, acute kidney injury before ICU admission, kidney transplant, morbidity obesity and limb amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients who developed acute kidney injury after ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Proportion of survivors in patients with AKI diagnosis during ICU | Up to 12 weeks after AKI diagnosis
  Patients admitted in ICU will be followed up to 2 weeks after AKI diagnosis and survival will be analyzed according to their hydration status assessed by BIVA.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Gonzalez, MD, PhD, Study Chair — Catholic University of Pelotas

IPD SHARING:
Plan to Share IPD: No